CLINICAL TRIAL: NCT05065892
Title: A Post-marketing Clinical Study of the Inactivated SARS-CoV-2 Vaccine (Vero Cells) (Produced in Wuhan): Immunogenicity and Safety Assessments in Patients With Hypertension and/or Diabetes
Brief Title: Evaluation of Immunogenicity and Safety of COVID-19 Vaccine (Produced in Wuhan) in Patients With Hypertension and/or Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Guizhou Center for Disease Control and Prevention (Other); Hunan Provincial Center for Disease Control and Prevention (Other); Center for Disease Control and Prevention, Fujian (Other); Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COVAX (HT/DM)-Wuhan
Record Dates: First submitted 2021-09-28; First posted 2021-10-04 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Serum testing technicians will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypertension group (Experimental): Hypertension group will enroll 330 subjects with hypertension (aged 60 years or older).
  Interventions: Biological: COVAX
- Diabetes Mellitus group (Experimental): Diabetes group will enroll 330 subjects with diabetes (aged 60 years or older).
  Interventions: Biological: COVAX
- Combined Disease group (Experimental): Combined Diseases group will enroll 300 subjects with both hypertension and diabetes (aged 60 years or older).
  Interventions: Biological: COVAX
- Healthy people group (Active Comparator): Healthy people group will enroll 480 subjects with no medical history of hypertension or diabetes (aged 60 years or older).
  Interventions: Biological: COVAX

INTERVENTIONS:
Biological: COVAX — 2 doses of Covid-19 vaccine

SUMMARY:
To evaluate the post-marketing immunogenicity and safety of the inactivated severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine (Vero cells) in patients aged 60 years or older with hypertension and/or diabetes, thus to further collect the immunogenicity and safety data of this product in special populations.

DETAILED DESCRIPTION:
After giving informed consent, patients with hypertension, patients with diabetes, patients with both diseases, and healthy controls, all aged 60 years or older, were given two doses of the inactivated SARS-CoV-2 vaccine (Vero cells). Venous blood samples were collected before the first dose and on day 28 after the second dose to evaluate the immunogenicity of the vaccine. Adverse events were actively recorded on a diary card once daily from day 0 to day 7 and once from day 8 to day 21 after the first dose and the second dose. Within 3 months after immunization with the second dose and collection of diary cards, the subjects were followed up by phone once a month as well as self-report to collect serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years old individuals with full civil capacity.
* Clinically confirmed body temperature of <37.3°C before enrolling in this study.
* Able and willing to participate in the study plan during the entire study and follow-up period.
* Capable of understanding the study procedures, willing to sign the informed consent form, and able to comply with the requirements of the clinical study protocol.
* Inclusion criteria for patients with hypertension and/or diabetes: Hypertension and/or diabetes definitively diagnosed by a community-level or higher medical institution. Patients with hypertension: systolic pressure <160 mmHg and diastolic pressure <100 mmHg on the day of immunization achieved by lifestyle adjustment and/or drug treatment; patients with diabetes: fasting glucose ≤13.9 mmol/L on the day of (or within 3 days before) immunization achieved by lifestyle adjustment and/or drug treatment.

Exclusion Criteria:

* Previously confirmed or asymptomatic COVID-19 patient.
* Has been immunized with a SARS-CoV-2 vaccine.
* Illiterate.
* Known allergy to any ingredient (including excipient) of this product.
* Received non-specific immunoglobulin injection within 1 month before enrollment.
* Received a live attenuated vaccine within 1 month before immunization or other vaccine within 14 days before immunization.
* Previous serious allergy to vaccine (e.g., acute allergic reaction, urticaria, angioedema, and dyspnea).
* Has uncontrolled epilepsy and other progressive neurological disorders; history of Guillain-Barré syndrome.
* Severe respiratory disorders, severe hepatic and renal diseases, malignancies, and various acute diseases or acute onset of chronic diseases.
* Diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases.
* Definitively diagnosed with thrombocytopenia or history of other coagulation disorders that may cause subcutaneous injection to be contraindicated.
* Currently experiencing acute complications (ketoacidosis, hyperosmolar state, lactic acidosis, etc.) of diabetes; or within 2 weeks after recovery from these complications.
* Other physical conditions judged by the investigator that render the patient unsuitable for participation in the clinical study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | Up to 28 days after the second dose
  the rate of positive seroconversion against coronavirus
Neutralizing antibody level | Up to 28 days after the second dose
  neutralizing antibody level against coronavirus

SECONDARY OUTCOMES:
Adverse events following vaccination | up to 6 months
  analyse the incidence of adverse events following immunization, both solicited and unsolicited

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nan'an Center for Disease Control and Prevention, Quanzhou, Fujian
  - Songtao Miao Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou
  - You County Center for Disease Control and Prevention, Zhuzhou, Hunan

IPD SHARING:
Plan to Share IPD: No